CLINICAL TRIAL: NCT02934763
Title: Opioid Induced Hyperalgesia (OIH) Modulation With Propranolol, in Laparoscopic Abdominal Surgery
Brief Title: Opioid Induced Hyperalgesia (OIH) Modulation With Propranolol
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-145
Record Dates: First submitted 2016-09-12; First posted 2016-10-17 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Hyperalgesia
MeSH Terms: conditions — Hyperalgesia | interventions — Propranolol; Adrenergic beta-Antagonists; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Saline solution by target controlled infusion
  Interventions: Drug: Saline
- Propranolol at 5ng/ml target dose (Active Comparator): Propranolol iv by target controlled infusion, to achieve a plasmatic concentration of 5ng/ml
  Interventions: Drug: Propranolol
- Propranolol at 15ng/ml target dose (Active Comparator): Propranolol iv by target controlled infusion, to achieve a plasmatic concentration of 15ng/ml
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — propranolol iv by target controlled infusion, to achieve specific plasmatic concentration goals
  Other Names: Beta blocker
  Arms: Propranolol at 15ng/ml target dose; Propranolol at 5ng/ml target dose
Drug: Saline — Saline as placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Opioid Induced Hyperalgesia (OIH) is an entity than has been demonstrated in healthy volunteers and in animal models. Is defined as an increase in the perception to painful stimuli, increasing the opioid requirements and diminishing the pain thresholds to stimuli.

The apparition of OIH is also related to the exposure to opioids during surgery, depending of the dose, the time of exposition and the type of opioid.

This condition can be modulated, specially in the perioperative context. It has been seen in healthy volunteers and in animal models, than the use of propranolol can modulate this phenomena, diminishing the postoperative requirements of analgesia. It is also unknown, the dose of propranolol required to modulate adequately OIH.

The objective of this work is to evaluate the efficacy of propranolol in the modulation of opioid induced hyperalgesia, with lower postoperative requirements of analgesia rescue.

DETAILED DESCRIPTION:
This is a randomized controlled study, comparing 2 interventions with a placebo. The interventions will be use of propranolol, at different doses, to achieve specific plasmatic concentrations.

80 patients will be required to find a difference of 20% in the primary outcome.

The primary outcome to be measured is the postoperative use of opioids in the post anesthesic care unit.

Secondary outcomes, will be the amount of opioids used in the following 24 hours to the surgery, the time to the first dose of analgesia in the post anesthesic care unit, and the change in the pain thresholds, evaluated as pain by pressure and by tactile sensitivity, before and after surgery.

Also, as a secondary outcome, in a group than will not receive the study drug, we will evaluate the temporal changes in opioid induced hyperalgesia, by pain sensitivity measured in the postoperative hours 2, 4 and 24. 10 patients receiving placebo will be part of this additional measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic cholecystectomy
* American Society of Anesthesiology Score (ASA) I-II

Exclusion Criteria:

* Medical history of cardiac disease
* Medical history of respiratory disease
* Regular use of beta blockers
* Known allergies to drugs used in the study
* Known history of illicit drugs use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid use | 24 hours posterior to surgery
  Dose of opioid required to manage pain adequately

SECONDARY OUTCOMES:
Pain thresholds (heat) | 24 hours posterior to surgery
  Evaluation of the threshold to perceive a heat perception as pain
Pain thresholds (cold) | 24 hours posterior to surgery
  Evaluation of the threshold to perceive a cold perception as pain
Pain thresholds (tactile sensitivity) | 24 hours posterior to surgery
  Evaluation of pain by tactile sensitivity, using the PinPrick system
Temporal changes in pain sensibility | 24 hours posterior to surgery
  Evaluation of pain by tactile sensitivity, using the PinPrick system

IPD SHARING:
Plan to Share IPD: Undecided